CLINICAL TRIAL: NCT04227145
Title: A Quasi-experimental, Interrupted Time Series Study to Evaluate the Effectiveness of "SexHealth Mobile" on Uptake of Contraception in Women With Substance Use Disorder
Brief Title: SexHealth Mobile: Integrating a Mobile Clinic and a Point-of-care Contraception Counseling and Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Swope Health Services (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001099
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-08

CONDITIONS: Contraceptive Usage; Contraception
Keywords: contraception; sexhealth mobile; substance abuse
MeSH Terms: conditions — Contraception Behavior; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): We will recruit up to 85 women with substance abuse disorder (or opioid abuse disorder) from recovery centers. Eligible women will complete a baseline survey and study staff will provide a referral for participants to seek more information on contraception and services. Study staff will record whether the participant accepted the referral. Follow-up will occur via phone call at 2-weeks, 1-month and 3-months post-enrollment to determine if they accessed contraceptive referral services if they initiated any contraceptive method, and if so: if they continued, changed, or discontinued this contraception method. We will recruit, complete baseline and usual care referral at recovery sites on a timely rotation that mirrors the intervention period (e.g., every fourth Friday morning at Site 1), in order to increase the chance of recruiting a comparable population.
- SexHealth Mobile (Experimental): We will train Swope providers in contraceptive counseling before intervention. We will recruit up to 85 women with substance abuse disorder (or opioid abuse disorder) from recovery centers. Eligible women will complete a baseline survey. Study staff will provide a referral for participants to seek more information on contraception and services. Women will have direct access to contraceptive counseling and services on-site via the mobile medical unit if they choose to use it. Counseling will focus on presenting the most effective contraceptive methods first (i.e., LARC). If women participate in contraceptive counseling, study staff will record the uptake of contraceptive medication and clinic referral at the time of enrollment and conduct follow-up surveys at 2-weeks, 1-month, and 3-months post-enrollment. If the participant refuses contraceptive counseling on MMU, a referral will be given.
  Interventions: Behavioral: SexHealth Mobile

INTERVENTIONS:
Behavioral: SexHealth Mobile — It will integrate two existing services in our community: a mobile medical unit (MMU) operated by Swope Health Services, and "SexHealth" a point-of-care contraception counseling service that our research team developed for Children's Mercy Hospital's emergency department (ED). Using a menu of adaptive services, "SexHealth Mobile" will bring contraceptive care to women with SUD (including a subset of women with OUD), if they wish to receive it, at targeted recovery sites Swope currently partners with.
  Arms: SexHealth Mobile

SUMMARY:
Pilot study aims to evaluate the effectiveness of "SexHealth Mobile" and improve access to highly effective contraception among women with substance use disorder (SUD) with "SexHealth Mobile" intervention. This intervention will consist of two existing services that will help reach women with or recovering from SUD and provide access to contraception, as well as counseling.

DETAILED DESCRIPTION:
Pilot study aims to evaluate the effectiveness of "SexHealth Mobile" and improve access to highly effective contraception among women with substance use disorder (SUD) with "SexHealth Mobile." Our study will follow a quasi-experimental design that uses an interrupted time series (i.e., usual care [control] then intervention care) to compare the uptake of contraception before and after implementing the "SexHealth Mobile" intervention.

"SexHealth Mobile" integrates two existing services in our community: a mobile medical unit (MMU) operated by Swope Health Services and "SexHealth" a point-of-care contraception counseling service that our research team developed for Children's Mercy Hospital's emergency department (ED) for adolescents. Using a menu of adaptive services, "SexHealth Mobile" will bring contraceptive care to women with SUD (including the subset with opioid use disorder [OUD]) at recovery centers in the Kansas City community.

Our primary hypothesis is that the current use of highly effective contraception will be greater at 1-month post-enrollment among women recruited during the intervention period (i.e., "SexHealth Mobile") compared to those recruited during the usual care period. The current use and discontinuation of contraception will also be compared at 2-weeks and 3-months.

Our approach consists of enrolling (n=170) eligible women are accessing health, recovery, or community services at a site we identified in our formative research work. We will aim to recruit up to 85 women during the usual care period and 85 during the intervention period. We will follow-up with participants at 2-weeks, 1-month, and 3-months after the enrollment date.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible if they:

* are between the ages of 18-40 years
* are biological females
* have an unmet need for contraception (sexually active, able to become pregnant, not consistently/currently using these contraception methods [sterilization, subdermal implant, intrauterine device, injectable, pill, patch, or ring]
* have current or recent (within the past year) problematic patterns of substance use (according to the CAGE-AID self-assessment

Exclusion Criteria:

Participants will be ineligible if they:

* have previously enrolled in the study
* are unable to provide informed consent
* are pregnant at index (recruitment) visit

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Miller, MD, Principal Investigator — Children's Mercy Emergency Department; Emily Hurley, PhD, Principal Investigator — Children's Mercy Health Services and Outcomes Research
Locations (4):
- United States (4):
  - Swope Health Services, Kansas City, Missouri
  - Amethyst Place: Swope Health Services Partner, Kansas City, Missouri
  - ReDiscover: Swope Health Services Partner, Kansas City, Missouri
  - Healing House Inc.: Swope Health Services Partner, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
After analysis, we will draft a de-identified results summary to be given to all partnering sites to share with their staff and clients.
Supporting Information: CSR

REFERENCES:
- [Result] Miller MK, Champassak S, Goggin K, Kelly P, Dowd MD, Mollen CJ, Humiston SG, Linebarger J, Apodaca T. Brief Behavioral Intervention to Improve Adolescent Sexual Health: A Feasibility Study in the Emergency Department. Pediatr Emerg Care. 2016 Jan;32(1):17-9. doi: 10.1097/PEC.0000000000000285. PMID 26727196
- [Result] Heil SH, Jones HE, Arria A, Kaltenbach K, Coyle M, Fischer G, Stine S, Selby P, Martin PR. Unintended pregnancy in opioid-abusing women. J Subst Abuse Treat. 2011 Mar;40(2):199-202. doi: 10.1016/j.jsat.2010.08.011. Epub 2010 Oct 30. PMID 21036512
- [Result] Terplan M, Hand DJ, Hutchinson M, Salisbury-Afshar E, Heil SH. Contraceptive use and method choice among women with opioid and other substance use disorders: A systematic review. Prev Med. 2015 Nov;80:23-31. doi: 10.1016/j.ypmed.2015.04.008. Epub 2015 Apr 18. PMID 25900803
- [Result] Haight SC, Ko JY, Tong VT, Bohm MK, Callaghan WM. Opioid Use Disorder Documented at Delivery Hospitalization - United States, 1999-2014. MMWR Morb Mortal Wkly Rep. 2018 Aug 10;67(31):845-849. doi: 10.15585/mmwr.mm6731a1. PMID 30091969
- [Derived] Hurley EA, Goggin K, Pina-Brugman K, Noel-MacDonnell JR, Allen A, Finocchario-Kessler S, Miller MK. Contraception use among individuals with substance use disorder increases tenfold with patient-centered, mobile services: a quasi-experimental study. Harm Reduct J. 2023 Mar 6;20(1):28. doi: 10.1186/s12954-023-00760-7. PMID 36879314

RESULTS

PARTICIPANT FLOW:
Period: Baseline and Post-Intervention Surveys
Arm/Group | Usual Care | SexHealth Mobile
Started | 48 | 50
Completed | 48 | 50
Not Completed | 0 | 0
Period: Two-week Follow-up
Arm/Group | Usual Care | SexHealth Mobile
Started | 38 | 31
Completed | 38 | 31
Not Completed | 0 | 0
Period: One-month Follow-up
Arm/Group | Usual Care | SexHealth Mobile
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0
Period: Three-month Follow-up
Arm/Group | Usual Care | SexHealth Mobile
Started | 36 | 22
Completed | 36 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | SexHealth Mobile | Total
Number analyzed (Participants) | 48 | 50 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 50 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 34] | 32.5 [28 to 35] | 31 [26 to 34]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 48 | 50 | 98
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 45 | 46 | 91
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 40 | 38 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 8 | 9
Region of Enrollment [Number; unit: participants]
  United States | 48 | 50 | 98
Contraception use [Count of Participants; unit: Participants] — Current use of hormonal contraception (pills, transdermal patch, vaginal ring, injection, subdermal implant) or intrauterine device. (Non-use was an eligibility criteria)
  Participants | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Current Use of Highly Effective Contraception
Description: Participants will be asked if they acquired birth control and their current use of it at 1-month period following the recruitment visit.
  Did participant initiate hormonal contraception or contraceptive device at initial visit or referral? Yes/No
  If yes, which contraception or contraceptive device was initiated? Implant/Depo-Provera/Birth control patch/Birth control pills/Birth control ring/Emergency contraception/ Intrauterine device
  If participant started using hormonal contraception or contraceptive device at 2-week follow-up time, are they still using hormonal contraception or contraceptive device at 1-month? Yes/No
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | SexHealth Mobile
Number analyzed (Participants) | 37 | 33
Participants | 2 | 17

2. Secondary Outcome: Current Use of Highly Effective Contraception
Description: Participants will be asked if they acquired birth control and their current use of it at 2-weeks and 3-months after recruitment visit
  Did participant initiate hormonal contraception or contraceptive device at initial visit or referral? Yes/No
  If yes, which contraception or contraceptive device was initiated? Implant/Depo-Provera/Birth control patch/Birth control pills/Birth control ring/Emergency contraception/ Intrauterine device
  If participant started using hormonal contraception or contraceptive device at 2-week follow-up time, are they still using hormonal contraception or contraceptive device at 3-month? Yes/No
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | SexHealth Mobile
Number analyzed (Participants) | 36 | 22
Participants | 5 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Usual Care | SexHealth Mobile
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT04227145/Prot_SAP_000.pdf